CLINICAL TRIAL: NCT04060485
Title: Screening Gene Mutations in Myeloid Cancers by Next Generation Sequencing to Improve Treatment Results
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201803002RIPD
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Aplastic Anemia
Keywords: Next generation sequencing; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Aplastic Anemia; Genetic mutation; Prognosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood or marrow blood will be obtained from routine practice blood/marrow sampling specimens (no extra venipuncture or bone marrow aspiration would be required).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic mutations have closely linked to the pathogenesis and prognostication of myeloid cancers. In addition, a number of molecularly targeted agents have been developed in recent years. With the advent of next generation sequencing (NGS), we now are able to detect a wide range of mutations more rapidly, accurately, and economically. In this study, the investigators will use NGS to screen and analyze myeloid-associated gene mutations in the participants, and aim to build up the mutational landscapes of the various myeloid cancers, and investigate how these mutations are linked to clinical outcome.

DETAILED DESCRIPTION:
Genetic mutations have closely linked to the pathogenesis and prognostication of myeloid cancers (including acute myeloid leukemia, myelodysplastic syndromes, and myeloproliferative neoplasms). In recent years, a number of novel therapeutic agents targeting various genetic mutations have been developed. For instance, patients with FLT3-ITD and IDH2 mutations have been shown to derive benefits from midostaurin and enasidenib, respectively. Furthermore, the TP53-mutated patients once categorized in the very high risk group, have been found to respond favorably to the hypomethylating agent, decitabine. Detecting a wide array of cancer mutations nowadays by the traditional Sanger method has become not only time-consuming but also not as cost-effective. With the advent of next generation sequencing (NGS), we now are able to detect a panel gene mutations more rapidly, accurately, and economically.

In this study, the investigators will screen and analyze myeloid-associated gene mutations in participants with myeloid cancers, with an in-house designed targeted NGS panel. The total nucleic acid from patients' blood or bone marrow specimens will be extracted, and then subjected to the library preparation procedure based on multiplex PCR amplification. Sequencing will be performed on Illumina MiSeq sequencer, and the results will be analyzed using our in-house developed bioinformatic workflow. Briefly, the sequenced reads will be aligned to human reference genome hg19 with BWA-mem, and somatic mutations called with Mutect2. The variants will be annotated via SnpEff with RefSeq, dbSNP, 1000 Genome Project, COSMIC and ClinVar databases. The investigators aim to build up the mutational landscapes of the above mentioned myeloid cancers, and investigate how these mutations are linked to clinical outcome.

ELIGIBILITY:
Inclusion criteria:

1. Patients ≥ 18 years of age diagnosed with myeloid cancers (including acute myeloid leukemia, myelodysplastic syndromes, and myeloproliferative neoplasms).
2. Healthy Volunteers ≥ 18 years of age.
3. Participants must be willing to provide voluntary written informed consent before study related procedures.

Exclusion criteria:

1. Patients ≥ 18 years of age diagnosed with non-myeloid cancers.
2. Patients <18 years of age diagnosed with myeloid cancers (including acute myeloid leukemia, myelodysplastic syndromes, and myeloproliferative neoplasms).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult myeloid cancer (including acute myeloid leukemia, myelodysplastic syndromes, and myeloproliferative neoplasms) patients (newly diagnosed or relapsed) diagnosed at the National Taiwan University Hospital (NTUH) according to the updated 2016 WHO myeloid disease classification.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-19 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of various genetic mutations in myeloid cancers | 5 years
  Peripheral blood or marrow blood will be obtained from routine practice blood/marrow sampling specimens (no extra venipuncture or bone marrow aspiration would be required) and sent for NGS analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chien Chou, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing and collaboration possibilities will be discussed upon request.